CLINICAL TRIAL: NCT00001991
Title: A Treatment IND for 566C80 Therapy of Pneumocystis Carinii Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 107A; 566-501
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-04

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: Trimethoprim-Sulfamethoxazole Combination; Pneumonia, Pneumocystis carinii; Antifungal Agents; Acquired Immunodeficiency Syndrome; atovaquone
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Atovaquone

INTERVENTIONS:
Drug: Atovaquone

SUMMARY:
To facilitate provision of atovaquone (566C80) to patients who have mild to moderate Pneumocystis carinii pneumonia (PCP) and are intolerant and/or unresponsive to trimethoprim / sulfamethoxazole (TMP / SMX ); to monitor serious adverse events attributable to 566C80.

ELIGIBILITY:
Inclusion Criteria

Patients must have the following:

* Clinical diagnosis of acute mild to moderate Pneumocystis carinii pneumonia.
* Dose-limiting intolerance to TMP / SMX or inadequate response to TMP / SMX.
* Willingness and ability to give informed consent. The clinical condition of the patient and appropriate physiologic criteria should be used in evaluating patients for therapy with 566C80. Patients who are rapidly progressing in disease severity or have severe disease as evidenced by sustained tachypnea (e.g., sustained respiratory rate > 30 breaths/minute), rapid deterioration in (A-a)DO2 and chest radiograph may not be appropriate candidates for oral therapy, including 566C80. Therapy with parenteral pentamidine should be undertaken in these cases. Treatment with IV trimetrexate or primaquine / clindamycin should be considered for these patients unless the patient is known to have dose-limiting intolerance to these agents. Patients with severe PCP who are intolerant and/or unresponsive to therapy with TMP / SMX and parenteral pentamidine may enroll in the 566C80 open-label compassionate plea protocol.

Exclusion Criteria

Patients with the following prior conditions are excluded: History of serious or dose-limiting adverse experience during previous 566C80 therapy, thought to be attributable to the drug.

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Glaxo Wellcome Inc, Research Triangle Park, North Carolina, United States